CLINICAL TRIAL: NCT03799315
Title: Reducing Tobacco-Related Health Disparities Among Incarcerated Individuals in Hennepin County
Brief Title: Jail-Based Use of Smoking Cessation Treatment Study
Acronym: JUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Hennepin County Adult Detention Center (Unknown); Brown University (Other)
Responsible Party: Principal Investigator, Tyler Winkelman, Clinician-Investigator, Hennepin Healthcare Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC-2018-0013
Record Dates: First submitted 2019-01-04; First posted 2019-01-10 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Tobacco Use
Keywords: Incarceration; Smoking; Counseling; Nicotine Replacement; Disparities
MeSH Terms: conditions — Tobacco Use; Smoking | interventions — Nicotine Replacement Therapy; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jail-Based Use of Smoking Cessation Treatment (JUST) (Experimental): Participants will receive guidline-based smoking cessation counseling while in jail and phone-based smoking cessation counseling sessions and nicotine lozenges after release from jail.
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: Counseling
- Enhanced Treatment As Usual (TAU) (No Intervention): Participants will receive the usual, limited smoking cessation treatment while in jail, plus an additional health and wellness education session in jail. Nicotine lozenges will be offered at the end of the study to those who did not quit smoking.

INTERVENTIONS:
Drug: Nicotine Replacement Therapy — All participants randomized to the JUST group will receive training on proper use of nicotine lozenges to aid in smoking cessation. Upon release from jail, participants will receive 2mg nicotine lozenges.
  Arms: Jail-Based Use of Smoking Cessation Treatment (JUST)
Behavioral: Counseling — All participants randomized to the JUST group will receive one hour of in-person, individual, guideline-based smoking cessation counseling during their jail stay. Upon release from jail, they will receive four 30-minute counseling phone calls over 3 weeks. These phone calls will take place at 24 hours, day 7, day 14, and day 20.
  Arms: Jail-Based Use of Smoking Cessation Treatment (JUST)

SUMMARY:
Smoking rates remain above 60% for individuals involved in the criminal justice system and contribute to elevated mortality rates in this population. Addressing smoking disparities among justice-involved individuals is a critical public health issue in Minnesota, one of a few states with rising incarceration rates. People who are incarcerated represent the intersection of multiple high-priority populations (disproportionately African-American, Native American, low-income, homeless, on Medicaid, and suffering from mental illness and substance use disorders). This study examines the impact of a smoking cessation intervention for individuals discharged from jail to the community on smoking abstinence. Participants will be randomized to either 1) guideline-based, in-person smoking cessation counseling during incarceration, telephone counseling after incarceration, and nicotine replacement, or 2) enhanced treatment as usual. This study's findings will be used to develop a larger, multi-site study that is fully powered to measure longer-term health and smoking cessation outcomes.

DETAILED DESCRIPTION:
Outcome assessments will be conducted for both arms at 1 week, 3 weeks, and 12 weeks post discharge from jail. During these assessments, seven-day point prevalence abstinence will be bio-verified with exhaled carbon monoxide, and self-reported general health, physical health, mental health, and substance use measures will also be obtained. The analysis is fully powered (i.e., power > .8) to detect significant between group effects on the primary outcome (i.e., the longitudinal, between group effect on bio-verified seven-day point prevalence abstinence over the 3 weeks post discharge). All analyses will be conducted on the intent to treat sample and will utilize pre-specified logistic and linear regression models.

ELIGIBILITY:
Inclusion Criteria:

* Use of ≥ 1 cigarette per day prior to incarceration
* Expected release from the Hennepin Adult Detention Center to the community within 90 days
* Age 18-64
* English fluency
* Lives within 20 minutes of Hennepin County Medical Center and has no plans to move away from area for 4 months
* Willing to attempt quitting or reducing smoking at discharge
* Has a telephone
* Cleared for nicotine lozenge safety by jail health care provider and willing to use at discharge

Exclusion Criteria:

* Active tuberculosis
* Current mental health crisis (i.e., currently experiencing significant mania, psychosis, or suicidality)
* Unable to ambulate independently
* Acute medical condition that would impair participant's ability to follow-up for assessments
* Expected discharge to a control institutional setting (e.g., locked state mental health facility or prison)
* Active pregnancy
* Heart attack within the last two weeks

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-08-29 (Actual)

PRIMARY OUTCOMES:
Bioverified 7-day point prevalence abstinence from smoking | Over 3 weeks
  Bioverified 7-day point prevalence abstinence from smoking

SECONDARY OUTCOMES:
Time to Lapse | 1 week, 3 weeks, 12 weeks
  Days to first lapse (i.e., any cigarette use, even a puff)
Time to Relapse | 3 weeks, 12 weeks
  Days to first relapse
Bio-verified 7-day point prevalence abstinence from smoking | Over 12 weeks
  Bioverified 7-day point prevalence abstinence from smoking
Health-related quality of life | 1 week, 3 weeks, 12 weeks
  Self-Reported health using the SF-12 total score and physical and mental health composite scores. Lower scores indicate worse health.
Depressive symptoms | 1 week, 3 weeks, 12 weeks
  The 10 item Center for Epidemiologic Studies Depression Scale (CESD-10) ranges from 0-30 with higher scores indicating higher depression symptoms.
Self-Reported Affect | 1 week, 3 weeks, 12 weeks
  10-item Positive and Negative Affect Scales (PANAS). The 5-item positive affect scale on the PANAS ranges from 5-25 with higher scores indicating greater positive affect. The 5-item negative affect scale on the PANAS ranges from 5-25 with higher scores indicating greater negative affect.
Health care utilization | 1 week, 3 weeks, 12 weeks
  Self-reported hospitalizations and use of the emergency department
Substance abuse | 1 week, 3 weeks, 12 weeks
  Self-reported substance abuse using the Drug Abuse Screening Test-10. Higher scores indicate more severe drug abuse.

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin Healthcare Research Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jamal A, King BA, Neff LJ, Whitmill J, Babb SD, Graffunder CM. Current Cigarette Smoking Among Adults - United States, 2005-2015. MMWR Morb Mortal Wkly Rep. 2016 Nov 11;65(44):1205-1211. doi: 10.15585/mmwr.mm6544a2. PMID 27832052
- [Background] Winkelman TNA, Vickery KD, Busch AM. Tobacco use among non-elderly adults with and without criminal justice involvement in the past year: United States, 2008-2016. Addict Sci Clin Pract. 2019 Jan 11;14(1):2. doi: 10.1186/s13722-019-0131-y. PMID 30635028
- [Background] Puljevic C, Kinner SA, de Andrade D. Extending smoking abstinence after release from smoke-free prisons: protocol for a randomised controlled trial. Health Justice. 2017 Dec;5(1):1. doi: 10.1186/s40352-016-0046-6. Epub 2017 Jan 23. PMID 28116579
- [Background] Binswanger IA, Carson EA, Krueger PM, Mueller SR, Steiner JF, Sabol WJ. Prison tobacco control policies and deaths from smoking in United States prisons: population based retrospective analysis. BMJ. 2014 Aug 5;349:g4542. doi: 10.1136/bmj.g4542. PMID 25097186
- [Background] Travis J, Western B, Redburn S, eds. The Growth of Incarceration in the United States: Exploring Causes and Consequences. Washington, D.C.: The National Academies Press; 2014. doi:10.17226/18613.
- [Background] Winkelman TN, Kieffer EC, Goold SD, Morenoff JD, Cross K, Ayanian JZ. Health Insurance Trends and Access to Behavioral Healthcare Among Justice-Involved Individuals-United States, 2008-2014. J Gen Intern Med. 2016 Dec;31(12):1523-1529. doi: 10.1007/s11606-016-3845-5. PMID 27638837
- [Background] Winkelman TN, Choi H, Davis MM. The Affordable Care Act, Insurance Coverage, and Health Care Utilization of Previously Incarcerated Young Men: 2008-2015. Am J Public Health. 2017 May;107(5):807-811. doi: 10.2105/AJPH.2017.303703. Epub 2017 Mar 21. PMID 28323472
- [Background] Vickery KD, Bodurtha P, Winkelman TNA, Hougham C, Owen R, Legler MS, Erickson E, Davis MM. Cross-Sector Service Use Among High Health Care Utilizers In Minnesota After Medicaid Expansion. Health Aff (Millwood). 2018 Jan;37(1):62-69. doi: 10.1377/hlthaff.2017.0991. PMID 29309230
- [Background] Frank JW, Linder JA, Becker WC, Fiellin DA, Wang EA. Increased hospital and emergency department utilization by individuals with recent criminal justice involvement: results of a national survey. J Gen Intern Med. 2014 Sep;29(9):1226-33. doi: 10.1007/s11606-014-2877-y. Epub 2014 May 10. PMID 24817280
- [Background] Clarke JG, Martin RA, Stein L, Lopes CE, Mello J, Friedmann P, Bock B. Working Inside for Smoking Elimination (Project W.I.S.E.) study design and rationale to prevent return to smoking after release from a smoke free prison. BMC Public Health. 2011 Oct 5;11:767. doi: 10.1186/1471-2458-11-767. PMID 21974746
- [Background] Clarke JG, Stein LA, Martin RA, Martin SA, Parker D, Lopes CE, McGovern AR, Simon R, Roberts M, Friedman P, Bock B. Forced smoking abstinence: not enough for smoking cessation. JAMA Intern Med. 2013 May 13;173(9):789-94. doi: 10.1001/jamainternmed.2013.197. PMID 23567902
- [Background] Mulder I, Tijhuis M, Smit HA, Kromhout D. Smoking cessation and quality of life: the effect of amount of smoking and time since quitting. Prev Med. 2001 Dec;33(6):653-60. doi: 10.1006/pmed.2001.0941. PMID 11716663
- [Background] Piper ME, Kenford S, Fiore MC, Baker TB. Smoking cessation and quality of life: changes in life satisfaction over 3 years following a quit attempt. Ann Behav Med. 2012 Apr;43(2):262-70. doi: 10.1007/s12160-011-9329-2. PMID 22160762
- [Background] Lemon SC, Friedmann PD, Stein MD. The impact of smoking cessation on drug abuse treatment outcome. Addict Behav. 2003 Sep;28(7):1323-31. doi: 10.1016/s0306-4603(02)00259-9. PMID 12915172
- [Background] Thurgood SL, McNeill A, Clark-Carter D, Brose LS. A Systematic Review of Smoking Cessation Interventions for Adults in Substance Abuse Treatment or Recovery. Nicotine Tob Res. 2016 May;18(5):993-1001. doi: 10.1093/ntr/ntv127. Epub 2015 Jun 11. PMID 26069036
- [Background] Busch AM, Tooley EM, Dunsiger S, Chattillion EA, Srour JF, Pagoto SL, Kahler CW, Borrelli B. Behavioral activation for smoking cessation and mood management following a cardiac event: results of a pilot randomized controlled trial. BMC Public Health. 2017 Apr 17;17(1):323. doi: 10.1186/s12889-017-4250-7. PMID 28415979
- [Background] A randomised controlled study of the Health Intervention "SNAP" in Northern Territory prisons- where smoking is banned- to prevent relapse to smoking. Trial Review. https://www.anzctr.org.au/Trial/Registration/TrialReview.aspx?id=371923. Published October 10, 2017. Accessed December 29, 2017.
- [Background] de Andrade D, Kinner SA. Systematic review of health and behavioural outcomes of smoking cessation interventions in prisons. Tob Control. 2016 Sep;26(5):495-501. doi: 10.1136/tobaccocontrol-2016-053297. Epub 2016 Oct 18. PMID 27798322
- [Background] Fiore MC, Jaen CR, Baker TB, et al. Treating Tobacco Use and Dependence: 2008 Update. Rockville, MD: U.S. Department of Health and Human Services. Public Health Service; 2008. https://bphc.hrsa.gov/buckets/treatingtobacco.pdf. Accessed October 17, 2017.
- [Background] Prisoner Research FAQs. HHS.gov. https://www.hhs.gov/ohrp/regulations-andpolicy/ guidance/faq/prisoner-research/index.html. Accessed December 18, 2017.
- [Background] Binswanger IA, Nowels C, Corsi KF, Long J, Booth RE, Kutner J, Steiner JF. "From the prison door right to the sidewalk, everything went downhill," a qualitative study of the health experiences of recently released inmates. Int J Law Psychiatry. 2011 Jul-Aug;34(4):249-55. doi: 10.1016/j.ijlp.2011.07.002. Epub 2011 Jul 29. PMID 21802731
- [Background] Wang EA, White MC, Jamison R, Goldenson J, Estes M, Tulsky JP. Discharge planning and continuity of health care: findings from the San Francisco County Jail. Am J Public Health. 2008 Dec;98(12):2182-4. doi: 10.2105/AJPH.2007.119669. Epub 2008 Apr 1. PMID 18381994
- [Background] Wang EA, Green J. Incarceration as a key variable in racial disparities of asthma prevalence. BMC Public Health. 2010 May 28;10:290. doi: 10.1186/1471-2458-10-290. PMID 20509891
- [Derived] Winkelman TNA, Ford BR, Dunsiger S, Chrastek M, Cameron S, Strother E, Bock BC, Busch AM. Feasibility and Acceptability of a Smoking Cessation Program for Individuals Released From an Urban, Pretrial Jail: A Pilot Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2115687. doi: 10.1001/jamanetworkopen.2021.15687. PMID 34228127